CLINICAL TRIAL: NCT01791777
Title: Effectiveness and Cost-effectiveness of Coaching Models to Promote Implementation of an Evidence-based Parenting Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); University of Georgia (Other)
Responsible Party: Principal Investigator, Daniel Whitaker, Director, National SafeCare Training and Research Center, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1R18CE001733 (NIH)
Record Dates: First submitted 2013-01-15; First posted 2013-02-15 (Estimated); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Child Maltreatment
Keywords: fidelity; implementation science; competence; training; coaching

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Purveyor (Experimental): The "purveyor" arm will include SafeCare Coaching that is conducted by a Training Specialists from the National SafeCare Training and Research Center (NSTRC), a GSU (Georgia State University)-Center that conducts training and research on the SafeCare model.
  Interventions: Behavioral: SafeCare Coaching
- Local (Experimental): The the "local" are will receive SafeCare Coaching that is provided by a staff member who works for the local social service agency.
  Interventions: Behavioral: SafeCare Coaching

INTERVENTIONS:
Behavioral: SafeCare Coaching — This study involves a comparison of different coaching models for providers who are newly trained to conduct an evidence-based parent training program (SafeCare). As part of all SafeCare trainings, all providers receive workshop training plus ongoing coaching to promote adherence to the intervention model. This research is aimed at understanding the coaching aspect of the training and dissemination processes, with the goal of implementing the most effective and efficient dissemination processes. One group of home visitors will be coached directly by NSTRC trainers, who work for NSTRC. The other group of home visitors will receive coaching that is provided by a staff member who works for the local social service agency.

SUMMARY:
The proposed study will compare purveyor coaching (conducted by National SafeCare Training and Research Center (NSTRC)) to local coaching that is supported by the purveyor (NSTRC). The outcomes of interest are home visitor fidelity and competence with the SafeCare model, and family engagement and skill acquisition. The study will also include a rigorous cost effectiveness analysis, and will examine individual and organizational factors that may affect implementation.

DETAILED DESCRIPTION:
This study is being conducted in the context of a nationwide implementation of SafeCare, an evidence-based parent training program. The primary goal of the research is to examine methods of coaching newly trained providers to implement a specific evidence-based practice. Thus, in this study, we are examining how two different coaching models affect provider fidelity and competence and parent's acquisition of the skills being trained. The primary participants in this study are the local coaches that will provide coaching to home visitors, the home visitors that will provide SafeCare to parents and the parents who will receive the SafeCare model. A total of 20 coaches, 90 home visitors and 270 parents have been proposed to participate in the study (n=380). The nature of participation in the study is similar for coaches and home visitors, but somewhat different for parents. Both groups will be asked to complete a variety of questionnaires at different time points, and allow observation of their performance with SafeCare delivery (for home visitors) and fidelity monitoring and coaching (for coaches). Observations may be done live or via audio recording. Parent participants will already be enrolled in SafeCare services, a voluntary parent-training program for parents, and will be invited to participate in this study by their home visitor. Parents' participation will involve completing a baseline and post-treatment in-home assessment before and after the SafeCare program, respectively. Each assessment will include an audio-computer assisted self-interview (ACASi), and an assessment of SafeCare skills. Parents will also complete 4 brief telephone interviews to assess their satisfaction and engagement with SafeCare services and provider competence. A more detailed list of data collection for coaches, home visitors, and trainers is as follows: Coaches: (1) prior to training/implementation, complete survey of individual and organizational variables that relate to implementation (2) allow observations of fidelity monitoring and coaching (3) report on home visitor competence, perceived self-competence, and support received from trainer (once per month for 6 months) (4) complete weekly time diaries reporting on time spent coaching (weekly for 6 months); Home visitors (1) prior to training/implementation, complete survey of individual and organizational variables that relate to implementation (2) allow and submit observations of SafeCare implementation (3) report on coach competence and support received from coach and perceived self-competence (once per month for 6 months); Families (1) complete baseline and post-treatment assessment involving behavioral observations and survey completed via ACASI (2) complete four short telephone interview reporting on home visitor competence and satisfaction with services.

ELIGIBILITY:
Inclusion Criteria:

* Providers administering SafeCare (Home Visitors and Coaches).
* Parents receiving SafeCare services from a Home Visitor how is also participating in the study.

Exclusion Criteria:

* Individuals under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in provider fidelity on the Home Visitor Fidelity Checklist. | Home Visitors will be monitored for the duration it takes up to five of their clients, who are also consented to participate in the study, to complete the SafeCare parent-training curriculum, an expected average of 6 months.
  As consistent with typical SafeCare implementation, the Home Visitors who provide the parent-training curriculum, SafeCare, to their clients will be monitored by a supervisor, their Coach, monthly to ensure fidelity to the SafeCare model is met. The Coach will listen to an audio recording the Home Visitor records of a session they have implementing SafeCare with their client and will grade the Home Visitor's performance using the Home Visitor Fidelity Checklist. The audio recording of the SafeCare session, the Coach's graded checklist of the session, as well as an audio recording the Coach captures of their feedback to the Home Visitor of the session and their checklist score will be captured every month.
Change in provider competency on the Home Visitor Competency Scale. | Home Visitors will be monitored for the duration it takes up to five of their clients, who are also consented to participate in the study, to complete the SafeCare parent-training curriculum, an expected average of 6 months.
  As consistent with typical SafeCare implementation, the Home Visitors who provide the parent-training curriculum, SafeCare, to their clients will be monitored by a supervisor, their Coach, monthly to ensure fidelity to the SafeCare model is met. The Coach will listen to an audio recording the Home Visitor records of a session they have implementing SafeCare with their client and will grade the Home Visitor's performance using the Home Visitor Fidelity Checklist. The audio recording of the SafeCare session, the Coach's graded checklist of the session, as well as an audio recording the Coach captures of their feedback to the Home Visitor of the session and their checklist score will be captured every month for purposes of fidelity monitoring. Blind coders will listen to the SafeCare sessions captured each month and score them using the Home Visitor Competency Scale.

SECONDARY OUTCOMES:
Time spent performing SafeCare coaching duties as recorded on the Time Diary form. | Coaches will record their time spent performing SafeCare coaching for the duration it takes up to five of their Home Visitor's clients to complete the SafeCare parent-training curriculum, an expected average of 6 months.
  SafeCare Coaches will record the time they spend performing SafeCare coaching duties every week on the Time Diary form. The form allows them to specify the date, number of minutes, content, and participating staff involved in each SafeCare activity they perform within the last week. Up to 26 weeks of Time Diaries will be collected to encompass the approximate 6-month study period.
Change in performance of parenting skills taught in the SafeCare parent-training program. | Time it takes SafeCare clients to complete the SafeCare parenting-training curriculum, approximately 4-6 months.
  Clients participating in the SafeCare parent-training curriculum will meet with their Home Visitors once a week for 18-20weeks and will be taught skills related to parent-child interactions, home safety, and identification and treatment of common child-illnesses. Home Visitors will assess client's use of the parenting skills before, during, and after the skills are taught to them; documents used to assess these skills will be collected by the research team. In addition, clients who participate in the study will complete two in-home assessments, once before starting the SafeCare program and once after completing the SafeCare program) which will involve data collection related to the three skill areas of SafeCare. Both the assessment documents collected by the Home Visitor during typical implementation as well as the data collected during the two in-home assessments will be used to determine the change in performance of clients who participate in the SafeCare parent-training program.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Whitaker, PhD, Principal Investigator — Georgia State Univeristy
Locations (10):
- United States (10):
  - Parent Aid Child Abuse Prevention Center, Tucson, Arizona
  - County of Humboldt - Department of Health and Human Services, Eureka, California
  - Family Support Services of North Florida Inc., Jacksonville, Florida
  - Georiga State University, Atlanta, Georgia
  - The Listening Ear, Conyers, Georgia
  - Pathways Transitions Programs, Decatur, Georgia
  - Children's Center of Surry, Inc., Dobson, North Carolina
  - Exchange Club of Durham North Carolina, Durham, North Carolina
  - Buckner Children & Family Services, Inc., Amarillo, Texas
  - Children's Connections, Inc., Lubbock, Texas

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data available.